CLINICAL TRIAL: NCT00584376
Title: A Multi-site, Double-blind, Randomized, Placebo-controlled, Crossover Study of Pregabalin (Lyrica, PGB) in the Treatment of Essential Tremor
Brief Title: Pregabalin (Lyrica) for the Treatment of Essential Tremor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Theresa Zesiewicz, Professor, University of South Florida
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Essential Tremor
Keywords: Essential tremor; tremor; pregabalin; lyrica
MeSH Terms: conditions — Essential Tremor; Tremor | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Pregabalin
  Interventions: Drug: Pregabalin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Gradually titrated dose ranging from 75mg po bid to 225mg po bid.
  Arms: 1
Drug: Placebo — Placebo capsules which are identical in packaging, appearance and dosing as the active capsules.
  Arms: 2

SUMMARY:
This will be a multi-site, prospective, double-blind, randomized, placebo-controlled, crossover trial conducted over 6 months to assess the effectiveness and safety of PGB to treat symptoms of ET.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients with essential tremor diagnosed by a movement disorder specialist.
2. Age 18 years to 80 years.
3. Postural tremor severity score of greater than or equal to 2 in the dominant hand/arm as measured by the FTM rating scale.
4. Women of child-bearing potential must use a reliable method of contraception and must provide a negative pregnancy test at entry into the study.
5. Baseline EKG read as within normal limits (no clinically significant abnormalities)obtained from primary care physician or cardiologist (performed within the past year).
6. Serum creatine kinase, complete metabolic blood count, liver function tests, renal function tests, and platelets are within normal limits (blood drawn within the past year).
7. Stable doses of all medications for 30 days prior to study entry and for the duration of the study.

Exclusion Criteria:

1. Any illness that in the investigator's opinion preclude participation in this study.
2. Pregnancy or lactation.
3. Concurrent participation in another clinical study.
4. Dementia or other psychiatric illness that prevents the patient from giving informed consent (Mini Mental Status Exam score less than 24).
5. Legal incapacity or limited legal capacity.
6. Presence of severe renal disease (BUN 50% greater than normal or creatine clearance <60 mL/min) or hepatic disease.
7. Presence of severe daytime sleepiness.
8. Abnormal creatine kinase and/or platelet count in the past year.
9. Present complaints of somnolence, dizziness, blurred vision, bleeding tendencies, cardiac abnormalities.
10. Previous lack of response to other ET therapies (propranolol AND primidone).
11. Patients who have had deep brain stimulation (DBS).
12. Concomitant treatment with gabapentin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Fahn-Tolosa-Marin Essential Tremor Rating Scale (FTM) total score | 61 days

SECONDARY OUTCOMES:
Writing tablet recordings of tremor amplitude | 61 days

CONTACTS AND LOCATIONS:
Overall Officials: Theresa A Zesiewicz, MD, Principal Investigator — University of South Florida
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Florida, Tampa, Florida
  - Emory Univ. School of Medicine, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Southern Illinois U. School of Medicine, Springfield, Illinois
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Vanderbilt, Nashville, Tennessee